CLINICAL TRIAL: NCT03354286
Title: Supporting Parents of Young Children With Type 1 Diabetes in Closed-Loop System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Colorado, Denver (Other); Indiana University (Other); Yale University (Other); University of South Florida (Other)
Responsible Party: Principal Investigator, Bruce A. Buckingham, Professor, Department of Pediatrics, Endocrinology and Diabetes Division, Stanford University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 43167
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: 670G; Hybrid closed-loop system; pediatric
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Growth and Development; Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Developmental & Technological Demands (Experimental): Provide education on using diabetes technology in various settings and formats in this age group, and increase ability for real-time problem-solving. Identify and troubleshoot barriers to keeping young children in Auto Mode.
  Interventions: Behavioral: Developmental & Technological Demands
- Distress Reduction (Experimental): Identify and reduce parent distress symptoms and worries. Provide strategies for obtaining social support.
  Interventions: Behavioral: Distress Reduction
- Nutrition, Set Point, & C:I Ratio (Experimental): Provide education on a variety of properties of food and how they affect blood glucose levels. Optimize the use of carbohydrate to Insulin ratios, insulin duration of action, and use of temporary target glucose set point in the 670G pump and the Quick bolus feature to gain better glycemic control.
  Interventions: Behavioral: Nutrition, Set Point, & C:I Ratio
- Hypoglycemia management (Experimental): Focus on hypoglycemia management to avoid hyperglycemia, review fear of hypoglycemia
  Interventions: Behavioral: Hypoglycemia management
- Minimal Intervention (Placebo Comparator): A short communication detailing the percentage of time spent in range and in Auto Mode and if the goals have been met.
  Interventions: Behavioral: Minimal Intervention

INTERVENTIONS:
Behavioral: Developmental & Technological Demands — Education and training related to use of CGM in this age group
  Arms: Developmental & Technological Demands
Behavioral: Distress Reduction — Education and training on reducing distress
  Arms: Distress Reduction
Behavioral: Nutrition, Set Point, & C:I Ratio — Education and training on how to use the HCL system to dose for different kinds of foods to improve glycemic control
  Arms: Nutrition, Set Point, & C:I Ratio
Behavioral: Hypoglycemia management — Education and training on reducing worries of hypoglycemia
  Arms: Hypoglycemia management
Behavioral: Minimal Intervention — Minimal intervention to simulate standard care - serves as the control group
  Arms: Minimal Intervention

SUMMARY:
This study will examine the impact of a closed-loop insulin delivery system intervention on health and psychological outcomes in families with young children with Type 1 Diabetes (T1D).

ELIGIBILITY:
To be eligible for the study, a child must meet the following criteria since enrollment in the CEP 302 Trial:

1. Diagnosis of type 1 diabetes according to ADA diagnostic criteria
2. Time since diagnosis of at least six months
3. Age between 2.00 and 6.99 years at enrollment
4. Parental consent to participate in the study
5. Completion of the CEP 302 Trial and in the continuation phase of the Medtronic CEP 302 Trial using the Medtronic MiniMed 670G pump with Enlite3 sensor.

To be eligible for the study, a parent must meet the following criteria:

1. Parent or legal guardian of a child with type 1 diabetes meeting the "child" criteria outlined above.
2. Age of 18.0 years or older.
3. Parent comprehends written English.
4. Parent understands the study protocol and signs the informed consent document.

The presence of any of the following is an exclusion for the study (since enrollment in the CEP 302 Trial):

1. Child has a medical disorder that in the judgment of the investigator will interfere with completion of any aspect of the protocol (e.g., pregnancy, kidney disease, adrenal insufficiency, skin condition that may hinder sensor application).
2. Child has a neurologic disorder that in the judgment of the investigator will affect completion of the protocol
3. Current use of oral glucocorticoids or other medications, which in the judgment of the investigator would be a contraindication to participation in the study
4. Child is unable to completely avoid acetaminophen for duration of study

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Time spent in blood glucose range | Change over 3 months
  Increasingly it is recognized that the percent time spent in a target blood glucose range, which is set by the American Diabetes Association, is an important outcome. This measure will be used as a primary outcome and derived from objective data downloads.

SECONDARY OUTCOMES:
Hemoglobin A1c | Change over 3 months
  The hemoglobin A1c value is a biologic measure of the glycemia that is the gold standard measure of "control" of diabetes. Collected through a blood sample.
Problem Areas in Diabetes | Change over 3 months
  This measure captures areas that are reported as problems for people with diabetes. Participants in the study report on daily problems with diabetes via this measure.
Parent Diabetes Distress Scale | Change over 3 months
  This measure is widely used to capture the psychological distress experienced in relation to diabetes.
Patient Health Questionnaire 8 | Change over 3 months
  This is a widely used measure that captures depressive symptoms. It is reported by the participants.
State-Trait Anxiety Inventory | Change over 3 months
  This is a widely used measure of anxiety symptoms. It is reported by the participant.
Pittsburgh Sleep Quality Index | Change over 3 months
  This questionnaire measures the degree to which sleep is disrupted and the quality of sleep experienced by participants.
Hypoglycemic Fear Survey - Parents | Change over 3 months
  People with diabetes worry about hypoglycemia. This measure captures those worries and is reported by participants.
Hypoglycemia Confidence Questionnaire | Change over 3 months
  Hypoglycemia needs to be managed in various daily situations. This questionnaire captures confidence of the participants in those various situations.
Pediatric Quality of Life Inventory | Change over 3 months
  This is a measure of health-related quality of life. It is used to understand the broader impact on quality of life which includes social, psychological, and health aspects of daily living.
Glucose Monitoring System Satisfaction Survey | Change over 3 months
  This a measure used to capture overall satisfaction with glucose monitoring devices used by participants.
General and diabetes-specific technology use | Change over 3 months
  This measure has questions on attitudes and use of various general technologies (e.g., smartphone) and diabetes devices.
Diabetes management behaviors | Change over 3 months
  Amount of time spent in Auto Mode; blood glucose monitoring frequency (by meter download); adherence to pump boluses. It is objectively reported by device downloads.
Health care utilization | Change over 3 months
  Number of visits and calls to the diabetes care team.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/86/NCT03354286/Prot_SAP_000.pdf